CLINICAL TRIAL: NCT00344721
Title: A Placebo Controlled Double Masked Clinical Assessment Study of Essential Fatty Acid Supplement and Its Effect on Patients With Apparent Aqueous Deficient Dry Eye Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Advanced Vision Research (Industry)
Responsible Party: Principal Investigator, James McCulley, Professor & Chairman, David Bruton Jr. Chair in Ophthalmology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 082004-008
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Dry Eye Syndrome
Keywords: Meibomian Gland Syndrome; Blepharitis
MeSH Terms: conditions — Dry Eye Syndromes; Blepharitis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either omega-3 fatty acid or placebo soft-gel capsules.
Who Masked: Participant, Outcomes Assessor
Masking Description: The active ingredient and placebo softgels appear identical and are supplied in identical containers for masking purposes.
  Study personnel performing study visit procedures are masked to group assignment.
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPA/DHA/flaxseed (Active Comparator): Study patients in the active comparator arm will take four soft-gel capsules containing omega-3 fatty acids (a nutritional supplement) orally daily for 3 months. Each daily dose contains eicosapentaenoic acid (450 mg), docosahexaenoic acid (300 mg) and flaxseed oil (1000 mg).
  Interventions: Dietary Supplement: Omega-3 fatty acid supplement
- Wheat germ oil (Placebo Comparator): Study patients in the placebo arm will take four doses of soft-gel capsules containing wheat germ oil orally daily for 3 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid supplement — Participants receive four oral doses of soft-gel capsules to be taken daily (QD) for 3 months.
  Arms: EPA/DHA/flaxseed
Dietary Supplement: Placebo — Participants receive four oral doses of soft-gel capsules containing wheat germ oil to be taken daily for 3 months.
  Arms: Wheat germ oil

SUMMARY:
To determine the effect of Essential Fatty Acids (EFA's) on Meibomian Gland lipids and aqueous tear production in patients with "dry eyes".

DETAILED DESCRIPTION:
The effects of essential fatty acids on Meibomian Gland lipid composition and aqueous tear production may be greater than previously thought. Dry Eye syndromes afflict millions of people worldwide, more than 10 million in the United States alone. Typically, symptoms that are associated with dry eye disease include ocular burning, foreign body sensation, photophobia and other symptoms that result in overall chronic discomfort in patients. Unfortunately, the effects of Essential Fatty Acids on aqueous tears or Meibomian lipids (AT) have not been established to date. The purpose of this study is to better understand the role essential fatty acids play in the maintenance of meibomian gland lipids and overall production or retention of aqueous tears.

Patients diagnosed with dry eye syndrome will be selected to participate in the study. Once qualified to take part in the trial, participants randomized to the active comparator arm will receive four oral doses of soft-gel capsules to be taken daily (QD). Omega-3 Fatty Acid daily content:

EPA (eicosapentaenoic acid) Dose: 450mg DHA (docosahexaenoic acid) Dose: 300mg Flaxseed Oil (organic) Dose: 1000mg

Patients on placebo will receive nutritional supplement capsules containing wheat germ oil but no EFA's. During the trial, patient will be encouraged not to change their diet, use of topical ophthalmics and systemic therapies other than the use of study treatment. Patient's topical therapy will be standardized after identification exam so that all patients will use TheraTears™ four times daily. Patients will be directed to take the masked capsules in the following manner: 4 soft-gels in the morning.

Masked medication, TheraTears™ and randomization tables will be provided by sponsor.

Subject will have the following tests performed during the first visit (before initiating treatment) and follow-up (after three months of treatment) visit,: a complete eye exam, (vital staining of ocular surface and tear break-up time); completion of questionnaires: Ocular Surface Index (OSDI) and Patient Symptomology Questionnaire will be presented to the patient to review and answer at both visits: Before initiating treatment and after three months on therapy, meibography, fluorophotometry will be performed in order to measure tear volume, flow and turnover, Schirmer test; and tear evaporation using an evaporimeter; meibomian gland drop out determined by infrared photography and meibomian gland secretion for biochemical analysis.

ELIGIBILITY:
Inclusion Criteria: Patient over 18 years of age, patient willing and able to comply with the protocol, no planned changes in diet, topical or systemic drugs during course of study. Ocular symptoms consistent with dry eye of insidious onset and greater than three months duration. Ocular surface vital staining consistent with aqueous deficient dry eyes with less than +1 conjunctival injection and no more than minimal lid inflammation -

Exclusion Criteria: Any patient that uses topical eye drops other than artificial tears. Any patient with punctual occlusion or punctual plugs. Patients with active ocular infection or inflammatory disease, history of herpetic keratitis, history of retinal detachment, concurrent contact lens use during the trial period, ocular surgery within the past six months, patients with glaucoma, anterior membrane dystrophy, active trichiasis or any eyelid globe malposition abnormality, e.g., entropion, ectropion, etc. Patients with Epiphora (excessive tearing). Moreover, patients taking medications known to effect aqueous tear production or meibomian secretions. Patient must not have participated in (or be currently participating in) any investigational therapeutic drug or device trial within the previous 30 days prior to their start date for this trial. In addition, any patient suffering from organic brain syndromes or major psychiatric disorder that would interfere with compliance or subjective reporting will be discouraged from participating in this trial.

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Lipid biochemistry changes: pre and post treatment | 3 months
  Meibomian gland secretions will be subjected to biochemical analysis.

SECONDARY OUTCOMES:
Evaporometry changes: pre and post treatment | 3 months
  Tear evaporation rate will be measured using an evaporometer.
Fluorophotometry changes:pre and post treatment | 3 months
  Clearance rate of the topically applied dye fluorescein will be measured by fluorophotometry.

CONTACTS AND LOCATIONS:
Overall Officials: James P. McCulley, M.D., Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No